CLINICAL TRIAL: NCT00609180
Title: Prospective, Randomized, Multi-Center Trial of Initial Trophic Enteral Feeding Followed by Advancement to Full-Calorie Enteral Feeding vs. Early Advancement to Full-Calorie Enteral Feeding in Patients With Acute Lung Injury (ALI) or Acute Respiratory Distress Syndrome (ARDS) and Prospective, Randomized, Blinded, Placebo-Controlled, Multi-Center Trial of Omega-3 Fatty Acid, Gamma-Linolenic Acid, and Anti-Oxidant Supplementation in the Management of Acute Lung Injury (ALI) or Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Early Versus Delayed Enteral Feeding and Omega-3 Fatty Acid/Antioxidant Supplementation for Treating People With Acute Lung Injury or Acute Respiratory Distress Syndrome (The EDEN-Omega Study)
Acronym: EDEN-Omega
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Omega arm of this study was stopped for futility. The EDEN arm continues to recruit patients as a separate independent study.
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 549; N01-HR056179, HSN268200536179C; N01HR056179 (NIH)
Record Dates: First submitted 2008-01-31; First posted 2008-02-06 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2012-02

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Acute Lung Injury; Acute Respiratory Distress Syndrome; Feeding; Critical Care; Ventilator; Omega-3 Fatty Acid; Antioxidant
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Participants will receive initial minimal (trophic) enteral feeding and the omega-3 fatty acid and anti-oxidant supplements
  Interventions: Behavioral: Minimal (Trophic) Feeding; Dietary Supplement: Omega-3 Fatty Acids and Antioxidant Supplements
- 2 (Experimental): Participants will receive initial full-calorie enteral feeding and the omega-3 fatty acid and anti-oxidant supplements
  Interventions: Behavioral: Full Feeding; Dietary Supplement: Omega-3 Fatty Acids and Antioxidant Supplements
- 3 (Experimental): Participants will receive initial minimal (trophic) enteral feeding and the placebo supplement
  Interventions: Behavioral: Minimal (Trophic) Feeding; Dietary Supplement: Placebo
- 4 (Placebo Comparator): Participants will receive initial full-calorie enteral feeding and the placebo supplement
  Interventions: Behavioral: Full Feeding; Dietary Supplement: Placebo

INTERVENTIONS:
Behavioral: Minimal (Trophic) Feeding — Enteral feeds will be started at 10 cc per hour and continued at this rate for 144 hours. After 144 hours of trophic enteral feeds, the feeding rate will be advanced to full-calorie rates, which will continue for the duration of mechanical ventilation up to Day 28.
  Arms: 1; 3
Behavioral: Full Feeding — Upon admission to the ICU, a full-calorie feeding rate will be determined, which will be calculated to deliver 25 to 35 kcal/kg predicted body weight (PBW) each day. Enteral feeds will be initiated at 25 cc per hour. The feeding rate will be increased by 25 cc per hour every 6 hours until goal rate is achieved, which will be administered for the duration of mechanical ventilation up to Day 28.
  Arms: 2; 4
Dietary Supplement: Omega-3 Fatty Acids and Antioxidant Supplements — Omega-3 fatty acids, GLA, and antioxidants will be administered through a feeding tube every 12 hours as a 120-cc bolus. Dosing will continue for 21 days or until discontinuation of mechanical ventilation.
  Arms: 1; 2
Dietary Supplement: Placebo — The study placebo will be administered through a feeding tube every 12 hours as a 120 cc bolus. Dosing will continue for 21 days or until discontinuation of mechanical ventilation.
  Other Names: TwoCal
  Arms: 3; 4

SUMMARY:
Acute respiratory distress syndrome (ARDS) and acute lung injury (ALI) are medical conditions that occur when there is severe inflammation and increased fluids in both lungs, making it difficult for the lungs to function properly. Hospital treatment for a person with ALI/ARDS often includes the use of a breathing machine, or ventilator, until the person is able to breathe without assistance. Initiating proper nutrition through a feeding tube early in a person's hospital stay may help to improve recovery, but the optimal timing, composition, and amount of feeding treatments are unknown. This study will evaluate whether early or delayed full-calorie feeding through a feeding tube is more effective in reducing recovery time and increasing survival rates in people with ALI/ARDS. The study will also determine whether supplementing the feedings with omega-3 fatty acids and antioxidants benefits people with ALI/ARDS.

DETAILED DESCRIPTION:
ALI/ARDS involves extensive inflammation in the lungs that can lead to rapid respiratory failure. These conditions are most commonly caused by pneumonia, generalized infection, or severe trauma to the lungs, but can also be less commonly caused by smoke or salt water inhalation, drug overdose, or shock.

For some people, ALI/ARDS resolves without treatment, but many severe cases result in hospitalization in the intensive care unit (ICU), where 30% to 40% of cases end in mortality. Current treatments for ALI/ARDS include assisted breathing with a ventilator, supportive care, and management of the underlying causes. Enteral feeding, in which patients receive nutrition through a feeding tube, plays an important role in treatment, too. Some recent studies have shown that, compared to delayed feeding, enteral feeding initiated soon after a patient begins assisted breathing is associated with a shorter hospital stay and a better chance of survival. However, other studies show the opposite, and studies on optimal feeding volume and composition have conflicting results. Studies have also indicated that enhancing enteral feeding with omega-3 fatty acid and antioxidant supplements may help reduce lung inflammation, improving overall recovery rates. This study will evaluate the effects of early versus delayed full-calorie enteral feeding on mortality, ventilator-free days, ICU-free days, and organ failure in people with ALI/ARDS. The study will also determine whether supplementation with omega-3 fatty acid and antioxidants adds any beneficial effect.

Upon admission to the ICU, a dietary evaluation will be done on each participant to determine goal, or full-calorie, feeding rates, which will be based on body weight and daily energy consumption. Participants will also undergo baseline assessments and procedures, which will include vital sign measurements, blood draws, a frontal chest radiograph, ventilator settings, and placement of feeding tube. Participants will be randomly assigned to receive initial enteral feedings that are either minimal (trophic) or full-calorie. They will also be randomly assigned to receive either omega-3 fatty acid and antioxidant supplementation or placebo. All participants will begin enteral feeding within 6 hours of treatment assignment.

Participants assigned to initial minimal enteral feedings will receive feedings at 10 cubic centimeters (cc) per hour, to be continued at this rate for 144 hours, provided that the participant remains on the ventilator. After the 144 hours, the feeding rate will be advanced to full-calorie rates.

Participants assigned to initial full-calorie enteral feedings will receive feedings at 25 cc per hour, and the feeding rate will be increased by 25 cc per hour every 6 hours until goal rate is reached. During enteral feedings, gastric residual volumes (GRVs) will be checked every 6 to 12 hours to assure acceptable levels. Participants will complete enteral feedings upon hospital discharge, Day 28 of treatment, death, or ability to achieve 48 hours of unassisted breathing. Omega-3 fatty acid, antioxidant, and placebo supplements will be administered with a syringe into the participant's feeding tube every 12 hours until Day 21 or discontinuation of the ventilator.

Blood pressure, heart rate, ventilation settings, and various blood factors will be measured during treatment. Phone-based follow-up assessments will occur at Months 6 and 12 after ICU discharge and will include measurements of health-related quality of life; psychological, neurocognitive, and physical activity outcomes; healthcare utilization; and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Must meet the following three criteria at study entry within a 24-hour period: 1) PaO2/FiO2 less than or equal to 300 (if altitude is more than 1000 meters, then PaO2/FiO2 less than or equal to 300 x [barometric pressure/760]), 2) bilateral infiltrates (patchy, diffuse, homogeneous, or asymmetric) consistent with pulmonary edema on frontal chest radiograph, and 3) requirement for positive pressure ventilation via endotracheal tube
* No clinical evidence of left-sided cardiac failure to account for bilateral pulmonary infiltrates
* Intention of primary medical team to enterally feed the patient
* Undergoes enteral feeding within 48 hours of meeting inclusion criteria

Exclusion Criteria:

* Neuromuscular disease that impairs ability to breath without assistance, such as cervical spinal cord injury at level C5 or higher, amyotrophic lateral sclerosis, Guillain-Barré syndrome, or myasthenia gravis
* Pregnant or breastfeeding
* Severe chronic respiratory disease. More information about this criterion can be found in the protocol.
* Burns on greater than 40% total body surface area
* Malignancy or other irreversible disease or condition for which 6-month mortality is estimated to be greater than 50%. More information about this criterion can be found in the protocol.
* Allogeneic bone marrow transplant within the 5 years before study entry
* Patient, surrogate, or physician not committed to full support (exception: a patient will not be excluded if he/she would receive all supportive care except for attempts at resuscitation from cardiac arrest)
* Severe chronic liver disease (Child-Pugh score of 11 to 15)
* Diffuse alveolar hemorrhage from vasculitis
* Morbid obesity, defined as 1 kg/cm body weight
* Unwilling or unable to use the ARDS network 6 mL/kg PBW ventilation protocol
* Moribund patient not expected to survive 24 hours
* No intent to obtain central venous access for monitoring intravascular pressures
* More than 72 hours since mechanical ventilation initiated
* Refractory shock. More information about this criterion can be found in the protocol.
* Unable to obtain enteral access
* Presence of partial or complete mechanical bowel obstruction
* Presence of ischemia or infarction
* Current total parenteral nutrition (TPN) use or intent to use TPN within 7 days of study entry
* Severe malnutrition with body mass index less than 18.5 or loss of more than 30% total body weight in the 6 months before study entry
* Laparotomy expected within 7 days of study entry
* Unable to raise head of bed 30 to 45 degrees
* Short-bowel syndrome or absence of gastrointestinal tract
* Presence of high-output (greater than 500 cc/day) enterocutaneous fistula
* International normalized ratio greater than 5.0, platelet count less than 30,000/mm3, or history of bleeding disorder
* Intracranial hemorrhage within the 1 month before study entry
* Allergy to enteral formula, omega-3 fatty acids, GLA, vitamin E, vitamin C, beta-carotene, taurine, or L-carnitine
* Requirement for, or physician insistence on, enteral formula supplemented with omega-3 fatty acids (ex: Oxepa®, Impact®) or providing omega-3 fatty acid, GLA, or antioxidant supplementation

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2007-12; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Number of ventilator-free days (VFD) | Measured at Day 28
Mortality before hospital discharge, with unassisted breathing | Measured at Days 60 and 90

SECONDARY OUTCOMES:
Number of intensive care unit-free days | Measured at Day 28
Number of organ failure-free days (liver, kidney, heart, central nervous system, and hematologic) | Measured at Day 28
Incidence of ventilator-associated pneumonia | Measured at Day 28
Number of days from first meeting criteria for weaning readiness to Day 28 | Measured at Day 28
VFDs and mortality in participants with a partial pressure of oxygen in arterial blood (PaO2)/fraction of inspired oxygen (FIO2) less than or equal to 200 or with shock at the time of study entry | Measured at Days 28 and 60, respectively
Change in plasma and mini-bronchoalveolar lavage (BAL) levels of interleukin (IL)-6, IL-8, von Willebrand factor (VWF), surfactant protein D (SPD), and total protein concentrations | Measured at Day 3
Health-related quality of life; healthcare utilization; and psychological, neurocognitive, and physical activity outcomes | Measured at Months 6 and 12
Duration of survival after hospital discharge using the National Death Index | Measured at Months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Wheeler, MD, Study Chair — Vanderbilt University Medical Center
Locations (41):
- United States (41):
  - University of San Francisco-Fresno Medical Center, Fresno, California
  - University of California, Davis Medical Center, Sacramento, California
  - UCSF-Moffitt Hospital, San Francisco, California
  - UCSF-San Francisco General Hospital, San Francisco, California
  - Centura St. Anthony Central Hospital, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Baton Rouge General Hospital-Blue Bonnet, Baton Rouge, Louisiana
  - Baton Rouge General Hospital-Midcity, Baton Rouge, Louisiana
  - Earl K. Long Medical Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Medical Center of Louisiana, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Baltimore VA Medical Center, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Maryland Shock Trauma Center, Baltimore, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - Rochester Methodist Hospital, Rochester, Minnesota
  - St. Mary's Hospital, Mayo Clinic, Rochester, Minnesota
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Durham Regional Medical Center, Durham, North Carolina
  - Moses Cone Health System, Greensboro, North Carolina
  - Wesley Long Community Hospital, Greensboro, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Harborview Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Brown SM, Wilson E, Presson AP, Zhang C, Dinglas VD, Greene T, Hopkins RO, Needham DM; with the National Institutes of Health NHLBI ARDS Network. Predictors of 6-month health utility outcomes in survivors of acute respiratory distress syndrome. Thorax. 2017 Apr;72(4):311-317. doi: 10.1136/thoraxjnl-2016-208560. Epub 2016 Jul 20. PMID 27440140
- [Derived] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Rice TW, Wheeler AP, Thompson BT, Steingrub J, Hite RD, Moss M, Morris A, Dong N, Rock P. Initial trophic vs full enteral feeding in patients with acute lung injury: the EDEN randomized trial. JAMA. 2012 Feb 22;307(8):795-803. doi: 10.1001/jama.2012.137. Epub 2012 Feb 5. PMID 22307571
- [Derived] Rice TW, Wheeler AP, Thompson BT, deBoisblanc BP, Steingrub J, Rock P; NIH NHLBI Acute Respiratory Distress Syndrome Network of Investigators. Enteral omega-3 fatty acid, gamma-linolenic acid, and antioxidant supplementation in acute lung injury. JAMA. 2011 Oct 12;306(14):1574-81. doi: 10.1001/jama.2011.1435. Epub 2011 Oct 5. PMID 21976613
- See also: Click Here for the NHLBI Acute Respiratory Distress Syndrome Network Website — http://www.ardsnet.org
- Available data/document: Individual Participant Data Set: ARDSNet-Omega — http://biolincc.nhlbi.nih.gov/studies/omega/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/omega/
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/omega/